CLINICAL TRIAL: NCT01791166
Title: Humoral Rejection - Diagnostic Markers in Pulmonary Transplant.
Brief Title: Immuno-humoral Rejection Markers in Pulmonary Transplant
Acronym: RHUM-TP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/49
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Lung Transplant
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary transplant (Experimental)
  Interventions: Biological: Blood test for detecting the circulatory anti-HLA antibodies by ELISA and LUMINEX tests

INTERVENTIONS:
Biological: Blood test for detecting the circulatory anti-HLA antibodies by ELISA and LUMINEX tests

SUMMARY:
Open multicentric prospective study performed on pulmonary transplanted patients to detect the values of different diagnostic markers for immuno- humoral reaction and their roles in the humoral rejection for those patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, more than 18 years of age.
* Patients with or without Cystic fibrosis
* Patients with no previous unilateral or bilateral pulmonary transplant or cardiopulmonary transplant
* Patients with no current other disease can affect, in short term, the process or prognosis of the transplant
* Patients had given his agreement to be enrolled in the study

Exclusion Criteria:

* Patient less than 18 year-old
* Patient had previous organ transplant
* Pregnant and/or lactating women
* Female subject in reproductive age does not use effective contraceptive methode
* Alcoholisms or neuropsychosis, conditions that affect the good comprehension of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of immune Markers of acute lung transplant rejection (Anti-HLA circulatory antibodies, neutrophils and C4d immune markers. | 12 months after pulmonary transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital FOCH, Suresnes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No